CLINICAL TRIAL: NCT06391528
Title: Effects of Transversalis Fascia Plane Block in Pediatric Patients Undergoing Inguinal Hernia and Orchiopexy Surgeries
Brief Title: Transversalis Fascia Plane Block in Pediatric Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, Principal Investigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024/06-19
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative; Regional Anesthesia; Parental Satisfaction
Keywords: postoperative pain; pain scores
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Control (No Intervention)
- Group FTB (Active Comparator)
  Interventions: Procedure: Transversalis Fascia Plane Block

INTERVENTIONS:
Procedure: Transversalis Fascia Plane Block — application of local anesthetic between the transversus abdominis muscle and the transversalis fascia surrounding it from the inside, at the level of the posterior axillary line.
  Arms: Group FTB

SUMMARY:
to investigate the effects of Transversalis Fascia Plan Block after induction of anesthesia on perioperative opioid consumption, hemodynamic changes, postoperative FLACC pediatric pain score, non-opioid analgesic use and parental satisfaction in pediatric patients undergoing unilateral inguinal hernia or undescended testicular repair under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 1-9 years old
* ASA I-II risk group
* Patients whose consent was obtained from their parents with an informed consent form
* Patients who will undergo Inguinal Hernia or Undescended Testi

Exclusion Criteria:

* ASA >2
* History of allergy to local anesthetics
* Known coagulation disorders
* Infection near the entry site
* Body mass index >30
* Those whose parents refused to participate in the study
* Those contraindicated for regional anesthesia
* Those with neurological or neuromuscular disease
* Patients with psychiatric problems
* Patients with a history of opioid use
* Chronic analgesic use
* Operation duration exceeding 2 hours

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain scores | up to 24 hour after surgery
  Patients will be evaluated at regular intervals after surgery and their pain will be measured using a FLACC scores.

SECONDARY OUTCOMES:
parental satisfaction | during the procedure
  asking parents about their satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University medicine faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No